CLINICAL TRIAL: NCT04367480
Title: Wireless Transcutaneous Electrical Nerve Stimulation (TENS) for Chemotherapy-Induced Peripheral Neuropathy: A Phase II Clinical Trial
Brief Title: Effects of Transcutaneous Electrical Nerve Stimulation on Chemotherapy-Induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester NCORP Research Base (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Gewandter, Assistant Professor, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: URCC19085; NCI-2019-07566 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); URCC19085 (Other: University of Rochester NCORP Research Base); URCC-19085 (Other: DCP); URCC-19085 (Other: CTEP); R21CA235389 (NIH); UG1CA189961 (NIH)
Record Dates: First submitted 2020-04-21; First posted 2020-04-29 (Actual); Results first posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group I (Active TENS) (Experimental): Patients wear an active wireless TENS device 5 hours daily for up to 6 weeks in the absence of unacceptable toxicity.
  Interventions: Other: Questionnaire Administration; Device: Transcutaneous Electrical Nerve Stimulation
- Group II (Placebo TENS) (Placebo Comparator): Patients wear a placebo wireless TENS device 5 hours daily for up to 6 weeks in the absence of unacceptable toxicity.
  Interventions: Device: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Device: Placebo Administration — Wear placebo TENS device
  Arms: Group II (Placebo TENS)
Other: Questionnaire Administration — Ancillary studies
Device: Transcutaneous Electrical Nerve Stimulation — Wear active TENS device
  Other Names: TENS; transcutaneous electric nerve stimulation
  Arms: Group I (Active TENS)

SUMMARY:
This phase II trial studies the effects of transcutaneous electrical nerve stimulation (TENS) for the treatment of peripheral neuropathy caused by chemotherapy, often called chemotherapy-induced peripheral neuropathy (CIPN). Peripheral neuropathy refers to the conditions that result when nerves that carry messages to and from the brain and spinal cord from and to the rest of the body are damaged or diseased. The TENS device emits high frequency electrical stimulation through the skin and may provide relief from chronic pain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Obtain efficacy estimates of daily TENS on CIPN (European Organization for Research and Treatment of Cancer-CIPN20 [EORTC-CIPN20]) to inform the design of a phase III confirmatory trial.

SECONDARY OBJECTIVES:

I. Obtain efficacy estimates of TENS on individual CIPN symptoms (i.e., hot/burning pain, sharp/shooting pain, tingling, numbness, cramping (measured daily via 0 - 10 numeric rating scale [NRS]).

II. Evaluate the feasibility of conducting, within the University of Rochester Cancer Center (URCC) National Cancer Institute Community Oncology Research Program (NCORP) network, a multisite, modified double-blind randomized control trial (RCT) of TENS for CIPN with physiologic assessments of descending inhibition (i.e., conditioned pain modulation [CPM] test) by assessing the proportions of (a) screened patients who enroll, (b) randomized participants who adhere to the treatment and complete the primary assessment, and (c) randomized participants who complete the CPM test.

EXPLORATORY OBJECTIVES:

I. Investigate the potential effects of TENS on balance, physical function, descending inhibition, lower limb sensation, and anxiety and depression.

II. Establish data to support the construct validity of the Treatment-Induced Neuropathy Assessment Scale (TNAS) and CIPN symptom inventory daily diary by comparison to the EORTC-CIPN20, which is the most commonly used measure of CIPN.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients wear an active wireless TENS device 5 hours daily for up to 6 weeks in the absence of unacceptable toxicity.

GROUP II: Patients wear a placebo wireless TENS device 5 hours daily for up to 6 weeks in the absence of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Have completed treatment with a platinum agent, taxane, vinca alkaloid, or bortezomib at least 3 months prior to registration
* Have a clinical diagnosis of CIPN from their physician or physician designee based on the following criteria: bilateral (i.e., present on both sides of the body), abnormal sensory symptoms in their feet or legs (e.g., hot/burning pain, sharp/shooting pain, numbness, tingling, cramping)
* Report at least 1 non-painful symptom associated with CIPN in their lower limbs (e.g., tingling, burning that isn't reported as painful, numbness)
* Report at least 2 of the following symptoms in their lower limbs (at their worst) as at least 4 out of 10 on a 0 - 10 NRS: hot/burning pain, sharp/shooting pain, numbness, tingling, cramping at visit 1 (i.e., week -1). Use the CIPN Symptom Inventory - week recall form (questions 1-5 ONLY) to assess these symptoms at screening
* Be willing and able not to start any new analgesic medications or change the dosages of any current analgesic medications (except acetaminophen [Tylenol] or non-steroidal anti-inflammatory drugs [NSAIDs] [i.e., ibuprofen (Advil, Motrin), naproxen (Aleve)]) for the duration of the study
* Be able to read English (i.e., is not illiterate, can speak English, and is not blind)
* Have access to a smart phone or device with an Apple or Android operating system that can be used to access the TENS device's application (App) and ability to connect to the internet on a daily basis during the trial

Exclusion Criteria:

* Have pre-existing neuropathy of any cause documented in their medical record prior to the start of chemotherapy or respond "yes" to the question "Did you have frequent numbness, tingling, sharp/shooting pain, hot/burning pain, or cramping in your feet before you started your chemotherapy?"
* Have unilateral CIPN symptoms (i.e., symptoms occur on predominantly only one side of the body)
* Be currently using a TENS device for any other reason
* Be currently taking, or have taken in the past 3 months, medications known to cause neuropathy in a significant portion of patients
* Have an acute and symptomatic lower extremity deep vein thrombosis (DVT) (treated DVT with resolution of symptoms is acceptable for enrollment)
* Lower extremity edema that is 2+ or greater (i.e., slight indentation that takes less than 15 seconds to rebound)
* Have started a new prescription pain medication or altered dosages of a prescription pain medication within the last 2 weeks
* Have lower extremity wounds or ulcers
* Have a cardiac pace maker or defibrillator
* Have epilepsy
* Have a leg that is too small or too large for the TENS device to fit securely
* Have missing lower limbs or amputations
* Have impaired decision making capacity (i.e., requires a legally authorized representative or health care proxy)
* Be pregnant or planning to get pregnant before expected completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Gewandter, Principal Investigator — University of Rochester NCORP Research Base
Locations (15):
- United States (15):
  - Christiana Health Care System, Newark, Delaware
  - Lee Memorial Health System, Fort Myers, Florida
  - Decatur Memorial Hospital, Decatur, Illinois
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Cancer Center at St. Mary's, Green Bay, Wisconsin
  - Aspirus, Wausau, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 participants withdrew from the study before randomization to an arm for the following reasons: Became ineligible after registration, Lost to follow-up, Changed their mind.
Period: Overall Study
Arm/Group | Group I (Active TENS) | Group II (Placebo TENS)
Started | 72 | 72
Received Intervention and Completed Baseline Assessments | 72 | 70
Completed | 68 | 62
Not Completed | 4 | 10
Not completed — Adverse Event | 1 | 1
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — App glitch during the study | 1 | 0
Not completed — Device Distribution Error | 0 | 2
Not completed — Ineligible after Randomization | 0 | 1
Not completed — Other Medical Reasons | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Active TENS) | Group II (Placebo TENS) | Total
Number analyzed (Participants) | 72 | 70 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (8.6) | 63.3 (10.7) | 62.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 51 | 92
  Male | 31 | 19 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 66 | 67 | 133
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 7 | 15
  White | 60 | 60 | 120
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 2 | 2
Education level [Count of Participants; unit: Participants]
  Less than High School | 1 | 2 | 3
  High School Graduate | 27 | 26 | 53
  College Degree | 30 | 27 | 57
  Graduate Degree | 14 | 14 | 28
  Chose not to answer | 0 | 1 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] — BMI calculation formulae - For standard measures: (weight (lb) / [height (in)]^2 ) x 703, For metric measures: weight (kg) / [height (m)]^2
  kg/m^2 | 30 (5.8) | 32 (7.9) | 31 (7.0)
Cancer Type [Count of Participants; unit: Participants]
  Breast | 20 | 31 | 51
  GI | 29 | 20 | 49
  Hematologic | 9 | 5 | 14
  Gynecologic | 7 | 6 | 13
  Other | 7 | 8 | 15
Neurotoxic Chemo Class [Count of Participants; unit: Participants]
  Platinum | 31 | 22 | 53
  Taxane | 20 | 32 | 52
  Platinum and Taxane | 12 | 11 | 23
  Bortezomib | 3 | 4 | 7
  Vinca alkaloid | 6 | 1 | 7
Time since Neurotoxic Chemo [Median (Inter-Quartile Range); unit: days] | 303 [170 to 735] | 667 [349 to 1129] | 454 [191 to 956]

OUTCOME MEASURES:

1. Primary Outcome: Chemotherapy-induced Peripheral Neuropathy (CIPN) Symptoms
Description: Measured by the mean European Organization for Research and Treatment of Cancer-CIPN20 (EORTC-CIPN20). The effects of transcutaneous electrical nerve stimulation (TENS) on CIPN will be estimated using analysis of covariance (ANCOVA).
  A 20 -item patient self -report tool to assess symptoms and function in the sensory, motor and autonomic domains.
  Two items, Q49 and Q50, were excluded from the total score calculation. Q49 was relevant only for individuals who could drive, and Q50 was relevant only for men.
  0 - 72, a higher score indicates worse neuropathy
Time Frame: 6 weeks after the start of intervention
Population: Participants who completed the baseline assessment were included in the analysis (N=141) except one extreme outlier that was removed from the Active TENS group due to data discordance among similar measures at baseline.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Group I (Active TENS) | Group II (Placebo TENS)
Number analyzed (Participants) | 71 | 70
score on a scale | 32.32 (0.57) | 33.37 (0.59)
Statistical Analysis 1: Comparison: Group I (Active TENS) vs Group II (Placebo TENS); Missing data were accounted for using multiple imputation (MI) with the fully conditional specification (FCS) method. 100 replicates were imputed. ANCOVA analysis was applied within each replicate. SAS PROC MI and MIANALYZE were used to calculate the reported estimates. (N: Active TENS=71, Placebo TENS=70); Test type: Superiority; p = 0.199, ANCOVA; Mean Difference (Final Values) = 1.05, 95% CI 2-sided [-0.56 to 2.67], Standard Error of Mean 0.81

2. Secondary Outcome: Effect of TENS on Hot/Burning Pain
Description: Measured by the CIPN Symptom Inventory; numeric rating scale of 0-10. Higher score is worse. The effects of transcutaneous electrical nerve stimulation (TENS) on hot/burning pain will be estimated using analysis of covariance (ANCOVA) for 2 study populations: (1) Study Completers (N: Active TENS=67, Placebo TENS=62) and (2) participants who reported at least 4 out of 10 at baseline for Hot/Burning Pain. (N: Active TENS=22, Placebo TENS=22).
Time Frame: 6 weeks after the start of intervention
Population: All participants who completed the study were included in the analysis, except one who did not provide Hot/Burning pain data at post-intervention.
Measure: Least Squares Mean (Standard Error); unit: mean of a score on a scale
Arm/Group | Group I (Active TENS) | Group II (Placebo TENS)
Number analyzed (Participants) | 67 | 62
mean of a score on a scale
  Study Completers | 1.80 (0.26) | 2.17 (0.27)
  Sample with Baseline >=4: number analyzed (Participants) | 22 | 22
  Sample with Baseline >=4 | 3.32 (0.60) | 4.69 (0.60)
Statistical Analysis 1: Comparison: Group I (Active TENS) vs Group II (Placebo TENS); Analysis on the Study Completers (N: Active TENS=67, Placebo TENS=62); Test type: Superiority; p = 0.302, ANCOVA; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-0.34 to 1.08], Standard Error of Mean 0.36
Statistical Analysis 2: Comparison: Group I (Active TENS) vs Group II (Placebo TENS); Subgroup analysis on participants who reported at least 4 out of 10 at baseline for Hot/Burning Pain. (N: Active TENS=22, Placebo TENS=22); Test type: Superiority; p = 0.112, ANCOVA; Mean Difference (Final Values) = 1.37, 95% CI 2-sided [-0.33 to 3.08], Standard Error of Mean 0.85

3. Secondary Outcome: Effect of TENS on Sharp/Shooting Pain
Description: Measured by the CIPN Symptom Inventory; numeric rating scale of 0-10. Higher score is worse. The effects of transcutaneous electrical nerve stimulation (TENS) on sharp/shooting pain will be estimated using analysis of covariance (ANCOVA) for 2 study populations: (1) Study Completers (N: Active TENS=67, Placebo TENS=62) and (2) participants who reported at least 4 out of 10 at baseline for Sharp/Shooting Pain. (N: Active TENS=24, Placebo TENS=23)
Time Frame: 6 weeks after the start of intervention
Population: All participants who completed the study were included in the analysis, except one who did not provide Sharp/Shooting pain data at post-intervention.
Measure: Least Squares Mean (Standard Error); unit: mean of a score on a scale
Arm/Group | Group I (Active TENS) | Group II (Placebo TENS)
Number analyzed (Participants) | 67 | 62
mean of a score on a scale
  Study Completers | 1.71 (0.25) | 2.04 (0.26)
  Sample with Baseline >=4: number analyzed (Participants) | 24 | 23
  Sample with Baseline >=4 | 2.87 (0.55) | 4.08 (0.56)
Statistical Analysis 1: Comparison: Group I (Active TENS) vs Group II (Placebo TENS); Analysis on the Study Completers (N: Active TENS=67, Placebo TENS=62); Test type: Superiority; p = 0.351, ANCOVA; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-0.37 to 1.02], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: Group I (Active TENS) vs Group II (Placebo TENS); Subgroup analysis was performed on participants who reported at least 4 out of 10 at baseline for Sharp/Shooting Pain. (N: Active TENS=24, Placebo TENS=23); Test type: Superiority; p = 0.128, ANCOVA; Mean Difference (Final Values) = 1.21, 95% CI 2-sided [-0.36 to 2.79], Standard Error of Mean 0.78

4. Secondary Outcome: Effect of TENS on Numbness
Description: Measured by the CIPN Symptom Inventory; numeric rating scale of 0-10. Higher score is worse. The effects of transcutaneous electrical nerve stimulation (TENS) on numbness will be estimated using analysis of covariance (ANCOVA) for 2 study populations: (1) Study Completers (N: Active TENS=67, Placebo TENS=62) and (2) participants who reported at least 4 out of 10 at baseline for Numbness. (N: Active TENS=60, Placebo TENS=50)
Time Frame: 6 weeks after the start of intervention
Population: All participants who completed the study were included in the analysis, except one who did not provide Numbness data at post-intervention.
Measure: Least Squares Mean (Standard Error); unit: mean of a score on a scale
Arm/Group | Group I (Active TENS) | Group II (Placebo TENS)
Number analyzed (Participants) | 67 | 62
mean of a score on a scale
  Study Completers | 4.78 (0.27) | 5.30 (0.28)
  Sample with Baseline >=4: number analyzed (Participants) | 60 | 50
  Sample with Baseline >=4 | 5.30 (0.26) | 5.57 (0.29)
Statistical Analysis 1: Comparison: Group I (Active TENS) vs Group II (Placebo TENS); Analysis on the Study Completers (N: Active TENS=67, Placebo TENS=62); Test type: Superiority; p = 0.166, ANCOVA; Mean Difference (Final Values) = 0.53, 95% CI 2-sided [-0.22 to 1.27], Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: Group I (Active TENS) vs Group II (Placebo TENS); Subgroup analysis was performed on participants who reported at least 4 out of 10 at baseline for Numbness. (N: Active TENS=60, Placebo TENS=50); Test type: Superiority; p = 0.492, ANCOVA; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.51 to 1.05], Standard Error of Mean 0.39

5. Secondary Outcome: Effect of TENS on Tingling
Description: Measured by the CIPN Symptom Inventory; numeric rating scale of 0-10. Higher score is worse. The effects of transcutaneous electrical nerve stimulation (TENS) on tingling will be estimated using analysis of covariance (ANCOVA) for 2 study populations: (1) Study Completers (N: Active TENS=67, Placebo TENS=62) and (2) participants who reported at least 4 out of 10 at baseline for Tingling. (N: Active TENS=55, Placebo TENS=50)
Time Frame: 6 weeks after the start of intervention
Population: All participants who completed the study were included in the analysis, except one who did not provide Tingling pain data at post-intervention.
Measure: Least Squares Mean (Standard Error); unit: mean of a score on a scale
Arm/Group | Group I (Active TENS) | Group II (Placebo TENS)
Number analyzed (Participants) | 67 | 62
mean of a score on a scale
  Study Completers | 4.32 (0.27) | 4.51 (0.28)
  Sample with Baseline >=4: number analyzed (Participants) | 55 | 50
  Sample with Baseline >=4 | 4.86 (0.29) | 5.10 (0.31)
Statistical Analysis 1: Comparison: Group I (Active TENS) vs Group II (Placebo TENS); Analysis on the Study Completers (N: Active TENS=67, Placebo TENS=62); Test type: Superiority; p = 0.622, ANCOVA; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.56 to 0.94], Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: Group I (Active TENS) vs Group II (Placebo TENS); Subgroup analysis was performed on participants who reported at least 4 out of 10 at baseline for Tingling. (N: Active TENS=55, Placebo TENS=50); Test type: Superiority; p = 0.587, ANCOVA; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.61 to 1.08], Standard Error of Mean 0.43

6. Secondary Outcome: Effect of TENS on Cramping
Description: Measured by the CIPN Symptom Inventory; numeric rating scale of 0-10. Higher score is worse. The effects of transcutaneous electrical nerve stimulation (TENS) on cramping will be estimated using analysis of covariance (ANCOVA) for 2 study populations: (1) Study Completers (N: Active TENS=67, Placebo TENS=62) and (2) participants who reported at least 4 out of 10 at baseline for Cramping. (N: Active TENS=18, Placebo TENS=18)
Time Frame: 6 weeks after the start of intervention
Population: All participants who completed the study were included in the analysis, except one who did not provide Cramping pain data at post-intervention.
Measure: Least Squares Mean (Standard Error); unit: mean of a score on a scale
Arm/Group | Group I (Active TENS) | Group II (Placebo TENS)
Number analyzed (Participants) | 67 | 62
mean of a score on a scale
  Study Completers | 1.61 (0.24) | 2.25 (0.25)
  Sample with Baseline >=4: number analyzed (Participants) | 18 | 18
  Sample with Baseline >=4 | 2.92 (0.58) | 4.27 (0.58)
Statistical Analysis 1: Comparison: Group I (Active TENS) vs Group II (Placebo TENS); Analysis on the Study Completers (N: Active TENS=67, Placebo TENS=62); Test type: Superiority; p = 0.058, ANCOVA; Mean Difference (Final Values) = 0.64, 95% CI 2-sided [-0.02 to 1.31], Standard Error of Mean 0.34
Statistical Analysis 2: Comparison: Group I (Active TENS) vs Group II (Placebo TENS); Subgroup analysis was performed on participants who reported at least 4 out of 10 at baseline for Cramping. (N: Active TENS=18, Placebo TENS=18); Test type: Superiority; p = 0.110, ANCOVA; Mean Difference (Final Values) = 1.35, 95% CI 2-sided [-0.32 to 3.02], Standard Error of Mean 0.82

ADVERSE EVENTS:
Time Frame: The adverse event data were collected over the intervention period. i.e. 6 weeks.
Description: Adverse events were assessed by phone in weeks 1, 3, and 5 and at the Week 6 visit. At each participant visit and phone call, the site study staff assessed adverse events by asking participants if they have experienced any new symptoms since starting the experimental treatment. They asked specifically if any skin reactions have occurred.
Arm/Group | Group I (Active TENS) | Group II (Placebo TENS)
All-Cause Mortality (participants affected / at risk) | 1/72 | 0/70
Serious Adverse Events (participants affected / at risk) | 1/72 | 1/70
Other Adverse Events (participants affected / at risk) | 17/72 | 12/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Active TENS) (N=72) | Group II (Placebo TENS) (N=70)
Disease Progression (General disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Active TENS) (N=72) | Group II (Placebo TENS) (N=70)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dysesthesia (Nervous system disorders) | 3 (3) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Muscle cramp (Nervous system disorders) | 0 (0) | 1 (1)
Burning sensation in toes (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT04367480/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT04367480/ICF_001.pdf